CLINICAL TRIAL: NCT03346720
Title: Ethical Challenges Related to Consent Following Implementation of a New Data Sharing Policy
Brief Title: Ethical Challenges of Consent in Data Sharing
Acronym: Data Sharing
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: BE1601
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Data Sharing
Keywords: Data Sharing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants recruited into biomedical research: Participants recruited into biomedical research where data collected may be shared with the wider research community.
  Interventions: Other: Semi-structured interviews; Other: Focus group discussions (FGDs)
- Frontline research staff: Frontline research staff directly involved in obtaining consent from participants in the above studies e.g. study nurses, investigators
  Interventions: Other: Semi-structured interviews; Other: Focus group discussions (FGDs)
- Research related staff and other stakeholders: Research related staff and other stakeholders involved in the implementation of the data sharing policy e.g. study managers, data access committee members, ethics committee members, study nurses, investigators, research collaborators, data managers and other clinical trials support staff.
  Interventions: Other: Semi-structured interviews; Other: Focus group discussions (FGDs)
- Community advisory board members: Community advisory board members and other community members
  Interventions: Other: Semi-structured interviews; Other: Focus group discussions (FGDs)

INTERVENTIONS:
Other: Semi-structured interviews — These interviews will be conducted following an interview guide. Interviews will be conducted in English or Thai at a place convenient and familiar to the interviewee. It is estimated that each interview will last between 45 minutes to an hour.
Other: Focus group discussions (FGDs) — These will be conducted following an interview guide. FGDs will be conducted in English or Thai. In addition, a note taker will be present to take notes. FGDs will take place at a place convenient and familiar to the participants. It is estimated that each FGD will last between 1 to 1.5 hours. FGDs will typically consist of homogenous groups e.g. study nurses.

SUMMARY:
In recent years, Mahidol Oxford Tropical Medicine Research Unit (MORU) has coordinated some of the largest international studies involving many sites in low-income and hard-to-reach settings. It has been our policy for many years to support sharing of data across collaborative research networks in order to maximize their utility. However there is increasing support from research funders, regulatory agencies and journals for sharing individual-level data from genomic, medical and public health research beyond research collaborations. A number of potential advantages of sharing individual level data from clinical and public health research have been identified in the literature. These include maximizing the utility of data, allowing verification of research results, and minimizing the burdens and costs of unnecessary duplication of research. In low- and middle-income settings it may be particularly important to effectively share data to maximize its utility and enable timely responses to important public health issues such as resistance to antimalarial treatments. Many authors have called for data sharing to be carefully curated, to minimize potential harms including breaches of privacy, the publication of poor quality or biased secondary research, and insufficient acknowledgment of the contribution of researchers generating datasets. In low- and middle-income settings, the need for data sharing policies and processes to promote equitable use of data, including the development of sustainable capacity to both share and analyse datasets, has been recognized.

It is foreseeable that the impact of this policy will be significant both practically and ethically. In the practical sense, there have already been changes in our data management processes and resources, clinical trial agreements and negotiations with collaborators. Ethically, this policy has impact on the consent process which includes the increasing use of broad consent, the changes in the language of information sheets, study protocols and ethics application documents and the actual consent taking by research staff.

Now that that these new data-sharing mechanisms have been put in place there is a need to evaluate their impact on practice. The aim of this study is to identify and analyse ethical challenges related to consent following implementation of a new data sharing policy with the aim of refining the data sharing policy and its related consent processes

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Able to speak and understand Thai, English, Burmese or Karen

Exclusion Criteria:

* Lack of relevant experience or expertise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four groups of participants will be recruited.
  Group 1. Participants recruited into biomedical research where data collected may be shared with the wider research community.
  Group 2. Frontline research staff directly involved in obtaining consent from participants in the above studies e.g. study nurses, investigators.
  Group 3. Research related staff and other stakeholders involved in the implementation of the data sharing policy e.g. study managers, data access committee members, ethics committee members, study nurses, investigators, research collaborators, data managers and other clinical trials support staff.
  Group 4. Community advisory board members and other community members.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
The opinion of ethical challenges in consent process under a new data sharing policy | 1 year

SECONDARY OUTCOMES:
The opinion of participants recruited in primary research with information presented to potential participations in future research studies about data sharing | 1 year
The views of stakeholders with broad consent | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Thailand (3):
  - Shoklo Malaria Research Unit, Mae Sot, Mae Sot, Changwat Tak
  - Hospital for tropical diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok
  - Mahidol-Oxford Tropical Medicine Research Unit (MORU) Office, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be de-identified and may be shared with other groups of researchers in accordance with the current MORU Data Sharing Policy.